CLINICAL TRIAL: NCT00166881
Title: Phase II Trial of Consolidation or Salvage Chemotherapy by Using Weekly Docetaxel/Irinotecan After Cisplatin Plus Weekly 24-Hour Infusion of High-dose 5-Fluorouracil/Leucovorin for Non-resectable Gastric Cancers
Brief Title: Weekly Docetaxel/Irinotecan for Non-resectable Gastric Cancers After Cisplatin Plus 5-FU/Leucovorin
Acronym: P-HDFL-DI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 57M9
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2012-11

CONDITIONS: Gastric Cancer
Keywords: Combination, Chemotherapy, Inoperable Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A, 2, III (Experimental): Weekly Docetaxel-Irinotecan for Inoperable Gastric Cancers After P-HDFL
  Interventions: Drug: Docetaxel-Irinotecan

INTERVENTIONS:
Drug: Docetaxel-Irinotecan — Docetaxel-Irinotecan, weekly, days 1, 8, 15, repeated every 4 weeks
  Other Names: Docetaxel (taxotere); Irinotecan (campto, CPT-11)

SUMMARY:
In this study, the investigators will use P-HDFL, a regimen with high tumor remission rate (~ 60-70%) and with only modest treatment-associated toxicities, as induction chemotherapy for patients with non-resectable gastric cancer. For those patients who have achieved complete response (CR) or partial response (PR), DI will be used to "consolidate" the remission. For those patients who fail to achieve remission by P-HDFL, DI will be used as salvage chemotherapy. The efficacy and toxicities of DI in these two settings will be evaluated in this prospective study.

DETAILED DESCRIPTION:
1. To evaluate if weekly Docetaxel-Irinotecan,a potentially non-cross-resistant regimen,can prolong the overall survival (OS) or the duration of remission in those patients who have achieved CR or PR by P-HDFL regimen
2. To evaluate the efficacy of weekly Docetaxel-Irinotecan combination as salvage regimen for those patients who have either failed to achieve remission or have recurred from P-HDFL chemotherapy
3. To find out the optimal doses for docetaxel and irinotecan in a weekly dosing schedule for gastric cancer patients
4. To evaluate the toxicities of weekly Docetaxel-Irinotecan regimen in inoperable gastric cancers

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed gastric adenocarcinoma
2. Measurable or evaluable disease
3. No previous C/T
4. Age 16 ~ 75 years
5. Karnofsky Performance Status of 60%
6. 4 weeks after R/T
7. Adjuvant C/T: the last dosing of C/T 6 months before enrollment
8. WBC >= 4,000, platelets >= 100K, Creatinine <= 1.5mg/dl and proteinuria <1+, normal serum bil, transaminase <= 3.5x ULN, TG > 70mg/dl

Exclusion Criteria:

1. CNS metastasis
2. Patients receive concomitant anti-cancer C/T or R/T
3. Patients who are pregnant and with an expected life expectancy less than 3 months
4. Symptomatic heart disease, active infection, extensive liver disease, or liver cirrhosis

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2000-06; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Five years

SECONDARY OUTCOMES:
Objective response rates (CR, PR) | Confirmed objective response after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Lii Cheng, M.D.,Ph.D., Study Chair — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan